CLINICAL TRIAL: NCT06510166
Title: The Effect of Distraction Methods Used During Inhalation Therapy on Children's Fear and Anxiety: A Randomized Controlled Study
Brief Title: The Effect of Distraction Methods Used During Inhalation Therapy on Children's Fear and Anxiety
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Merve Koyun, Principal Investigator, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: OndokusMK
Record Dates: First submitted 2024-07-06; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Child; Inhalation Therapy; Complications; Fear; Distraction Methods; Anxiety
Keywords: child; inhalation theraphy; fear; distraction methods; anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- normal nebulizer + mask + distraction technique (Experimental): Inclusion criteria is below:
  1. Parent and child volunteer to participate in the study,
  2. The child is between 3-6 years old,
  3. Presentation due to upper and lower respiratory tract infection,
  4. Inhaler treatment will be applied with a nebulizer,
  5. No request for any other intravenous, intramuscular or invasive treatment,
  6. The child does not have any genetic, congenital, chronic or metabolic disease
  Interventions: Behavioral: Children's Fear and Anxiety normal nebulizer and mask+ distraction
- toy type nebulizer + toy mask (Active Comparator): Inclusion criteria is below:
  1. Parent and child volunteer to participate in the study,
  2. The child is between 3-6 years old,
  3. Presentation due to upper and lower respiratory tract infection,
  4. Inhaler treatment will be applied with a nebulizer,
  5. No request for any other intravenous, intramuscular or invasive treatment,
  6. The child does not have any genetic, congenital, chronic or metabolic disease
  Interventions: Behavioral: Children's Fear and Anxiety a toy nebulizer and a toy mask
- control group (No Intervention): Inclusion criteria is below:
  1. Parent and child volunteer to participate in the study,
  2. The child is between 3-6 years old,
  3. Presentation due to upper and lower respiratory tract infection,
  4. Inhaler treatment will be applied with a nebulizer,
  5. No request for any other intravenous, intramuscular or invasive treatment,
  6. The child does not have any genetic, congenital, chronic or metabolic disease

INTERVENTIONS:
Behavioral: Children's Fear and Anxiety normal nebulizer and mask+ distraction — Children in group 2 will receive their inhaler treatment with a normal nebulizer and mask, while at the same time one of the distraction techniques of their choice (drawing a picture, reading a story or watching an age-appropriate cartoon) will be applied.
  Arms: normal nebulizer + mask + distraction technique
Behavioral: Children's Fear and Anxiety a toy nebulizer and a toy mask — Children in Group 3 will receive their inhaler treatment using a toy nebulizer and a toy mask.
  Arms: toy type nebulizer + toy mask

SUMMARY:
It was aimed to examine the effects of distraction methods used during inhalation therapy on children's fear and anxiety.

Hypothesis:

Hypothesis 0 (H0): There is no difference between the fear and anxiety levels of children who received normal nebulizer + mask + distraction techniques and toy type nebulizer + toy mask during inhaler treatment and the children in the control group.

Hypothesis 1 (H1): The fear and anxiety levels of children who received normal nebulizer + mask + distraction techniques during inhaler treatment are lower than the children in the control group.

Hypothesis 2 (H2): The fear and anxiety levels of children who were applied a toy type nebulizer + toy mask during inhaler treatment are lower than the children in the control group.

Hypothesis 3 (H3): The fear and anxiety levels of children who were treated with a toy type nebulizer + toy mask during inhaler treatment were lower than those of children who were treated with a normal nebulizer + mask + distraction techniques.

DETAILED DESCRIPTION:
In the literature, distraction techniques are generally used in invasive procedures. On the other hand, it is possible that studies on the effects of inhalation therapy and non-pharmacological methods, which are among the common non-invasive interventions in children, can still continue. Durak et al. (2021) stated that the developments in experimental groups, in which they were made to watch cartoons during inhalation treatment, were lower in adults than in control groups and in children. A similar study was published by Ozsamuri (2020), and children receiving mask and inhaler treatment consisted of watching cartoons, listening to music, and a control group. As a result of the study, intra-group comparisons show that the fear and anxiety scores of people in cartoon and music groups decreased compared to before the procedure . However, arranging emergency services for children and selling them with treatment materials have been shown to be effective in reducing children's fears. Negative reactions to the growth mask and nebulizer during inhaler therapy, causing incorrect inhalation patterns, and deterioration are reduced. Yanık and Ayyıldız (2019) conducted a study on the effectiveness of the training given with a toy-type nebulizer for children aged 3-6 years who received nebulizer therapy. During the therapy inhaler treatment, the scores of the people in the experimental group decreased, while the scores of the control group increased. Kırkan (2023) stated that the therapeutic play method applied with toy nebulizers and toy nebulizers in the activities he conducted with 3-8 year old children who received nebulizers is an effective method treatment in reducing fear and anxiety in the children's hospital. Distracting methods during inhaler treatment for children are beneficial for patients to have positive hospital experiences. This will reduce patients' fear of the hospital, prevent providers from experiencing stress, and ensure that people are satisfied. Adequate information during treatment procedures in children will improve fear, pain and anxiety management and increase the positive hospital experience. Rapid healing is important because of the reduced use of treatment materials, the effectiveness of human resources, and the increase in health knowledge.

ELIGIBILITY:
Inclusion Criteria:

* Parent and child volunteer to participate in the study,
* The child is between 3-6 years old,
* Presentation due to upper and lower respiratory tract infection,
* Inhaler treatment will be applied with a nebulizer,
* No request for any other intravenous, intramuscular or invasive treatment,
* The child does not have any genetic, congenital, chronic or metabolic disease,

Exclusion Criteria:

* Parent and child are not willing to participate in the study,
* The child is not between 3-6 years old,
* Presentation for a reason other than upper and lower respiratory tract infection,
* No inhaler treatment with a nebulizer,
* Request for any other intravenous, intramuscular or invasive treatment,
* The child has any genetic, congenital, chronic or metabolic disease

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2024-10-08 (Estimated); Study Completion 2024-12-08 (Estimated)

PRIMARY OUTCOMES:
changing the anxiety | 'Before inhalation theraphy within 5 minutes', 'During inhalation theraphy' and 'After inhalation theraphy within 5 minutes'
  Children's Anxiety Meter- State (CAM-S) is designed like a thermometer, featuring a bulb at its base and horizontal markers at regular intervals as it ascends. Children are asked to represent their feelings on this scale by marking where they stand "right now". They are instructed, "Imagine that all your anxious or angry feelings are on the bulb or bottom part of the thermometer. If you are a little worried or nervous, the feelings may go up a little on the thermometer. If you are very, very anxious or nervous, emotions can go all the way to the top. Put a line on the thermometer showing how anxious or nervous you are." This scale provides scores ranging from 0 to 10. As the score increases, the level of anxiety increases.
changing the fear | 'Before inhalation theraphy within 5 minutes', 'During inhalation theraphy' and 'After inhalation theraphy within 5 minutes'
  Children's Anxiety Meter- State (CAM-S) is designed like a thermometer, featuring a bulb at its base and horizontal markers at regular intervals as it ascends. Children are asked to represent their feelings on this scale by marking where they stand "right now". They are instructed, "Imagine that all your anxious or angry feelings are on the bulb or bottom part of the thermometer. If you are a little worried or nervous, the feelings may go up a little on the thermometer. If you are very, very anxious or nervous, emotions can go all the way to the top. Put a line on the thermometer showing how anxious or nervous you are." This scale provides scores ranging from 0 to 10. As the score increases, the level of anxiety increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Ondokuz Mayıs University, Samsun, Atakum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
other researchers may view the study once it is published.

REFERENCES:
- [Background] Durak H, Uysal G. The Effect of Cartoon Watching and Distraction Card on Physiologic Parameters and Fear Levels During Inhalation Therapy in Children: A Randomized Controlled Study. J Trop Pediatr. 2021 Jan 29;67(1):fmab018. doi: 10.1093/tropej/fmab018. PMID 33742204
- [Background] Kirkan C, Kahraman A. Effect of therapeutic play using a toy nebulizer and toy mask on a child's fear and anxiety levels. J Pediatr Nurs. 2023 Nov-Dec;73:e556-e562. doi: 10.1016/j.pedn.2023.10.033. Epub 2023 Nov 7. PMID 37940393